CLINICAL TRIAL: NCT01715025
Title: An Open-labeled Pilot Study to Determine the Efficacy of an E2//Nomegestrol Acetate (E2/NOMAC)Combination Oral Contraceptive (COC) in the Management of Heavy Menstrual Bleeding (HMB)
Brief Title: A New Treatment Option for Heavy Menstrual Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sydney Centre for Reproductive Health Research (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2012-7
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Menorrhagia
Keywords: measured; heavy menstrual bleeding; combined oral contraceptive; alkaline haematin method
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E2/Nomac (Experimental): Women with demonstrated HMB at baseline will be assigned to 3 cycles of a E2/Nomac combined pill 1 daily for 24 days followed by 1 placebo pill daily for 4 days per cycle.
  Interventions: Drug: E2Nomac

INTERVENTIONS:
Drug: E2Nomac — Women will start the first cycle of the COC on the first day of their period in the treatment phase of the study
  Other Names: Zoely

SUMMARY:
Women with measured menstrual bleeding >80ml per cycle and no contraindications to combined oral contraceptive use will be assigned to an oestradiol/nomegestrol acetate oral contraceptive for 3 cycles during which they will collect all menstrual blood and send all used sanitary protection to the laboratory at the University of Sydney for estimation of blood loss by the alkaline haematin method.

Hypothesis:

An estradiol/nomogestrel acetate (E2/NOMAC) combined pill will be effective in controlling HMB in the majority of women without structural pelvic pathology.

Main outcome:

The primary efficacy end-point will be the proportion of women with a reduction of menstrual blood loss ≥ 50% from baseline.

DETAILED DESCRIPTION:
Women will collect menstrual blood for 3 cycles and will be eligible to enter the treatment phase if in two of the three pre-treatment cycles the measured menstrual blood loss (MBL)is >80ml. The mean of these baseline MBL measurements will be the comparator for the efficacy treatment measurement. Iron studies (serum ferritin, Fe and transferrin) will also be measured pre and post treatment and related to women's assessment of their quality of life measured on a validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 years having regular menstrual cycles
* Women willing to collect all sanitary protection for 6 cycles
* Women with no contraindications to use of combined hormonal contraception
* Women not using any hormonal contraception or any treatment for HMB
* Women who have no demonstrable uterine pathology on pelvic ultrasound
* Women who have demonstrated a menstrual blood loss (MBL) >80mls in 2 of 3 menstrual periods during the pre-treatment phase will be eligible to enter the treatment phase

Exclusion Criteria:

* Women for whom combined oral contraceptives are contraindicated
* Women unwilling to collect all sanitary protection for 6 cycles
* Women using hormonal contraception or any treatment for HMB
* Women who have demonstrable uterine pathology on pelvic ultrasound
* Women who have demonstrated a MBL ≤80mls in 2 of 3 consecutive menstrual periods

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
• The primary efficacy end-point will be the proportion of women with a reduction ≥ 50% from baseline | Baseline to outcome 12weeks
  A single arm open label intervention study

SECONDARY OUTCOMES:
•• A secondary efficacy endpoint will be the number and proportion of cycles with a normal blood loss ≤ 80mls | •Baseline to endpoint 12 weeks
  Open label single group measuring the efficacy of a combined hormonal contraceptive to restore a normal level of MBL

CONTACTS AND LOCATIONS:
Overall Officials: Edith Weisberg, MB BS MM, Principal Investigator — Sydney Centre for Reproductive Health Research FPNSW
Locations (1):
- SCRHR, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Fraser IS, Romer T, Parke S, Zeun S, Mellinger U, Machlitt A, Jensen JT. Effective treatment of heavy and/or prolonged menstrual bleeding with an oral contraceptive containing estradiol valerate and dienogest: a randomized, double-blind Phase III trial. Hum Reprod. 2011 Oct;26(10):2698-708. doi: 10.1093/humrep/der224. Epub 2011 Jul 21. PMID 21784734